CLINICAL TRIAL: NCT05334745
Title: Clinical Comparison of Topical Application of Alvogyl Versus Topical Application of Hyaluronic-Acid Gel in Management of Pain And Palatal Wound Healing : A Randomized Controlled Clinical Trial
Brief Title: Clinical Comparison of Topical Application of Alvogyl Versus Hyaluronic-Acid Gel in Management of Pain And Palatal Wound Healing
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, mohy eldin mahmoud aboelazayem, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01005007001
Record Dates: First submitted 2022-04-07; First posted 2022-04-19 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Wound Healing
MeSH Terms: interventions — butyl aminobenzoate, eugenol, iodoform, spearmint oil drug combinations; Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- application of Alvogyl in the palatal wound with stent (Experimental)
  Interventions: Other: Alvogyl
- application of 0.2% Hyaluronic acid is placed in the palatal wound with stent . (Other)
  Interventions: Other: Alvogyl

INTERVENTIONS:
Other: Alvogyl — application of Alvogyl in the palatal wound with stent versus hyaluronic acid application
  Other Names: Hyaluronic acid

SUMMARY:
The aim of the study is to evaluate the effect of application of Alvogyl versus hyaluronic acid in decreasing postoperative pain and promoting healing in the palatal wound following the free gingival graft procedure

DETAILED DESCRIPTION:
Postoperative pain and bleeding are the most common complications after palatal graft harvesting, also postsurgical swelling have been reported. Although hemostatic agents, mechanical barriers, bioactive materials, antibacterial and antiseptic agents and herbal products have been found effective in preventing such complications, an ideal support could not be specified for this purpose. Further, undesired side effects such as delayed wound healing/foreign body reaction have been reported .

No gold standard has been identified, thus there is a need for further investigations aiming to reach the best possible treatment modality for pain relief and prevention of reported complications following harvesting of palatal graft .

ELIGIBILITY:
Inclusion Criteria:

* Patients with mucogingival defects scheduled for free gingival graft
* Age from 18 years up to 60
* Medically healthy patient

Exclusion Criteria:

* Systemic diseases that may be a contraindication for any surgeries.
* Loss of maxillary premolars and molars.
* Pregnancy or lactation
* Smoking

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
postoperative pain | 7th days
  Pain through one week using the visual analogue scale (VAS)

SECONDARY OUTCOMES:
Wound healing | 7th, 14th, 21st and 30th days.
  * Wound healing index through one month .
  * The healing index has 5 grades which are 5(excellent healing), 4(very good healing), 3 (good healing), 2(poor healing) and 1(very poor healing)

CONTACTS AND LOCATIONS:
Locations (1):
- Egypt, Cairo, Egypt